CLINICAL TRIAL: NCT01283048
Title: A Phase I Study of Bevacizumab and Escalation Doses of BKM-120 in Patients With Metastatic Renal Cell Carcinoma Who Failed Prior Systemic Therapies
Brief Title: Bevacizumab and BKM-120 in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toni Choueiri, MD (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor-Investigator, Toni Choueiri, MD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-405
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney Cancer; Avastin
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM-120 Bevacizumab (Experimental): BKM-120 60, 80, 100 mg PO QD Bevacizumab 10 mg/Kg every 2 weeks
  Interventions: Drug: BKM-120 Bevacizumab

INTERVENTIONS:
Drug: BKM-120 Bevacizumab — BKM-120 60, 80, 100 mg PO QD Bevacizumab 10 mg/Kg every 2 weeks
  Other Names: Avastin

SUMMARY:
BKM-120 is a drug that may slow the growth of cancer cells. This drug has been used in laboratory experiments and information from those research studies suggests that this drug may help to slow the growth of renal cancer cells. In this research study, the investigators are testing the safety to BKM-120 at different dose levels. The investigators will also be studying how well tolerated BKM-120 is, and how effective BKM-120 can be in the treatment of kidney cancer.

DETAILED DESCRIPTION:
Subjects will receive an intravenous infusion of Avastin on Day 1 and Day 15 of each month (cycle). Subjects will take a daily oral dose of BKM-120 at the dose level assigned.

Subjects will have a clinic visit weekly during Cycle 1 and then on Day 1 and Day 15 of each cycle for blood tests and physical exam.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic RCC with clear cell component or papillary RCC
* Life expectancy > 12 weeks
* Must have failed at least 1 prior anti-VEGF systemic therapy for metastatic RCC

Exclusion Criteria:

* Prior treatment with a P13K inhibitor or bevacizumab
* Untreated brain metastases
* Acute or chronic liver or pancreatic disease
* Major mood disorder
* Concurrent severe and/or uncontrolled medical condition
* Diabetes mellitus
* GI disease
* Currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant
* Pregnant or breastfeeding
* HIV positive
* History of another malignancy within 3 years except cured basal cell carcinoma of the skin or excised in situ carcinoma of the cervix
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and dose limiting toxicities of the combination of BKM-120 and bevacizumab in metastatic renal cell carcinoma | 2 year

SECONDARY OUTCOMES:
To determine additional toxicity and safety information from the combination of BKM-120 and bevacizumab in an expanded cohort of patients at the MTD | 2 year
To determine the objective response proportion, progression-free survival, overall survival of the combination of BKM-120 and bevacizumab | 2 years
To determine whether the BKM-120 and bevacizumab combination at the MTD is associated with concomitant changes in angiokines and PI3K pathway members in plasma and tumor samples | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Toni K Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan